CLINICAL TRIAL: NCT07364968
Title: Evaluating the Impact of Randomized Preoperative Instructional Video on Patient Preparedness Following Minimally Invasive Gynecologic Surgery
Brief Title: Impact of a Preoperative Instructional Video on Patient Preparedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Sarah Simko, M.D., Principal Investigator, University of California, Riverside
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23031
Record Dates: First submitted 2025-10-24; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Laparoscopic Surgery; Minimally Invasive Surgical Procedures
Keywords: Minimally invasive surgical procedures

STUDY DESIGN:
Intervention Model Description: control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group of patients will be asked to watch an informational video. (Active Comparator): They will be encouraged to ask their provider any follow-up questions. A link to view the video an unlimited amount of times will be provided.
  Interventions: Other: Study group of patients will receive standard of care
- Study group of patients will receive standard of care (No Intervention): The group of patients will receive the standard patient education in place before the procedure and will also be able to ask to follow-up questions from their provider. All patients will receive a link to complete a preoperative questionnaire.

INTERVENTIONS:
Other: Study group of patients will receive standard of care — The group of patients will receive the standard patient education in place before the procedure and will also be able to ask to follow-up questions from their provider.
  Arms: Study group of patients will be asked to watch an informational video.

SUMMARY:
In this study, the investigators will evaluate the impact of a pre-operative instructional video for patients undergoing minimally invasive gynecologic surgery. The video will educate patients to understand what to expect and how to take care of themselves after the procedure. The effectiveness of the video will be evaluated via a questionnaire to see if patients who watched the video had better recovery outcomes, greater understanding, and less anxiety when compared to the group of patients who did not watch the pre-operative video.

The two questions the investigators wish to address are:

1. Will the patients who watch the pre-operative will show decreased anxiety and uncertainty about their procedure when compared to the control group?
2. Will increased understanding of the information shared in the video result in less pain medication usage, less ambiguity and thus increased compliance with post-operative care instructions, and quicker recovery?

DETAILED DESCRIPTION:
The study group of patients will be asked to watch the informational video about what to expect after their procedure and instructions on how to recover. They will be encouraged to ask their provider any follow-up questions. A link to view the video an unlimited amount of times will be provided. The control group of patients will receive the standard patient education in place before the procedure and will also be able to ask to follow-up questions from their provider. All patients will receive a link to complete a preoperative questionnaire.

Both groups will be scheduled for their routine two-week postoperative visit. At this visit, the questionnaire will be given to the patients in the form of a link to a virtual questionnaire to evaluate for effectiveness of the pre-operative video.

ELIGIBILITY:
Participants/Sample Size: Female patients who have been recommended for minimally invasive gynecologic surgery. A total of 52 patients will be enrolled in this study at UCR Women's Health Clinic. Statistical power: To detect an effect size of 0.5 with a power of 0.8, a sample size of 52 participants was required.

Inclusion criteria:

* Age 18 - 65 years old
* Surgery with UCR Gynecology physician
* Laparoscopic/robotic surgery
* Same day discharge after surgery
* Can read a survey in English
* Female

Exclusion Criteria:

* Receiving postoperative chemotherapy in the 6-week postoperative period
* Minors under the age of 18
* Postoperative overnight stay
* Laparotomy (open surgery)
* Pregnancy

Max Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
patient level of satisfaction with the education they received prior to surgery | 6 months to one year
  Our primary outcomes will be patient level of satisfaction with the education they received prior to surgery and its impact on post-operative care which will be measured by the standardized likert scale (1 to 5 scale where 1 = strongly disagree and 5= strongly agree). The survey will include the following objective and subjective measures: Tylenol tablets used (over two weeks), Ibuprofen tablets used (over two weeks), pain scale (1 to 5 scale where 1 = none and 5= very severe). Additional information will be collected from the patient's medical records (ie. office visit notes, telephone encounters, hospital laboratory results, pain medication refill requests). Patients should continue any medication regimen as instructed by their physician up to the day of surgery. Patients will be treated for complications as they would have been treated otherwise. Study duration period will be approximately six months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Riverside, California, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant-level data will not be released. Only data aggregated to remove any identifiers will be made available.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT07364968/Prot_SAP_000.pdf
  • Informed Consent Form: UCR Template Consent (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT07364968/ICF_001.pdf